CLINICAL TRIAL: NCT01826656
Title: A Clinical/Real Time Model of Intramembranous Jawbone Healing in Post-menopausal Osteoporotic and Non-osteoporotic Women. A Pilot Study.
Brief Title: Bone Healing in Healthy and Post-menopausal Osteoporotic Women
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit suitable patients
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OsteoporosisTrial
Record Dates: First submitted 2013-03-26; First posted 2013-04-08 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Post-menopausal Osteoporosis
Keywords: intramembranous bone healing; post-menopausal osteoporosis; tooth extraction
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Tooth Extraction; Absorptiometry, Photon; Radiography, Panoramic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- post-menopausal osteoporotic women (Other): Subjects of test group will follow a tooth extraction and they will perform a CBCT scan within 10 days from the extraction and after 3 months (+/-15 days)
  Interventions: Procedure: tooth extraction; Radiation: CBCT scan; Radiation: DXA scan; Radiation: Panoramic radiograph
- non-osteoporotic post-menopausal women (Active Comparator): Subjects of the control group will follow a tooth extraction and will perform a CBCT scan within 2 days from the extraction and after 3 months (+/- 2 days)
  Interventions: Procedure: tooth extraction; Radiation: CBCT scan; Radiation: DXA scan; Radiation: Panoramic radiograph

INTERVENTIONS:
Procedure: tooth extraction — Patients from both groups will follow the extraction of an hopeless tooth
Radiation: CBCT scan — A CBCT scan will be performed within 2 days from the tooth extraction at after 3 months (+/-2 days)
Radiation: DXA scan — DXA scan will be performed at the hip and lumbar spine in all self-reported non-osteoporotic subjects who hasn't done one within 1 year, to confirm their normal bone mineral density. Osteoporotic subjects already have a DXA scanner.
Radiation: Panoramic radiograph — As basic standard of care, a panoramic radiograph will be performed to both test and control subjects who haven't done one within the previous year, in order to give them a full-mouth dental diagnosis

SUMMARY:
Both the pathogenesis and the treatment of osteoporosis may potentially interfere at different levels on the multi-stage complex cascade of events involved in bone healing/regeneration. To our knowledge no human studies have been performed to clarify the potential effect of osteoporosis on post-extraction alveolar healing. The primary outcome of the study is to compare alveolar bone changes in width and height 3 months after tooth extraction in 10 post-menopausal osteoporotic women and 10 post menopausal non osteoporotic women by the use of cone-beam computer tomography (CBCT) images. The secondary outcomes considered are: clinical changes in the external contour of the ridge and periodontal parameters in the neighbouring teeth after a tooth extraction and 3 months later. In addition the accuracy of panoramic morphometric indexes in detecting osteoporosis will be measured.

DETAILED DESCRIPTION:
Despite some contradictory results, there is significant pre-clinical evidence, mainly deriving from fracture studies, of a delay in bone formation together with a decrease in bone mineral density and mechanical resistance in osteoporotic-like conditions. Very few human data are available, mainly deriving from retrospective speculations, but they seem to confirm the existence of a delay in consolidation subsequent to bone fractures, a higher rate of orthopedic complications and a reduction in mechanical strength. Some pre-clinical and clinical studies have also supported a negative effect of osteoporosis on bone graft healing and implant success, but controversial opinions exist.

A useful model to study the influence of osteoporosis on bone healing is the post-extraction socket healing, with consideration of the absence of cartilage formation, the short period needed to heal and its clinical relevance.

The animal studies reported controversial results, but a general reduction and a delay in bone formation with an increase in bone turnover was usually observed in ovariectomized rats. No human studies have clarified the effect of osteoporosis on post-extraction alveolar healing. This pilot study will try to shed light on this topic.

As there are no similar studies in the literature, we estimated that 10 post-menopausal osteoporotic women (test) and 10 healthy pre or post-menopausal women (control) would be a convenient sample to collect enough data for our purpose. This will also allow us to collect information about the variance to power a further study (if needed).

In this study, women who need the extraction of a single tooth due to fracture, destroying caries, periodontitis, endodontic or prosthetic reasons will be included. The tooth should present at least 30% of its periodontal attachment preserved. All the patients will be provided a full-mouth diagnosis of soft and hard tissues, detailed hygiene instructions and the careful removal of plaque and tartar in a highly controlled research environment as part of the project and all the treatment will be free of charge. Subjects of the test group will be recruited among newly diagnosed post-menopausal osteoporotic women attending the Rheumatology clinic at the University College of London Hospital, whilst subjects of the control group will be recruited among healthy women attending the Eastman Dental Institute. Written informed consent will be obtained prior to any clinical evaluation. Differences between test and control groups will be assessed at each time interval using either parametric (if data are normally distributed with approximately equal variances) or non-parametric tests.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian women, > 50 years old
* women referring to have reached a menopause status, defined as the permanent cessation of the ovulation, since at least 1 year and presenting a diagnosis of osteoporosis based on dual X-rays energy absorptiometry (DXA) measurement of the bone mineral density at the femur neck or lateral spine (t value 2.5 SD or more below the young female adult mean) (TEST GROUP)
* women in menopausal status since at least 1 year and with normal bone mineral density, as assessed by DXA scan (CONTROL GROUP)
* subjects needing a tooth extraction. The tooth to extract should present at least 30% of its attachment level preserved. Wisdom teeth are excluded from this study
* Subjects must have voluntarily signed the informed consent.

Exclusion Criteria:

* on hormone replacement therapy (HRT) or taking any other drugs (except Vit D and calcium) for the treatment of osteoporosis (e.g. biphosphonates)
* on chronic treatment (i.e., two weeks or more) with any medication known to affect oral status (e.g., phenytoin, cyclosporine, and non-steroidal anti-inflammatory drugs) within one month from baseline visit.
* affected by systemic diseases recognized to affect bone metabolism (e.g. Cushing's syndrome, Addison's disease, non-controlled diabetes mellitus, leukemia, pernicious anemia, malabsorption syndromes, chronic liver disease, rheumatoid arthritis..)
* on therapy with drugs that can affect bone metabolism (e.g. glucocorticoids, anticonvulsants, anticoagulants, benzodiazepines, cytotoxic drugs, immunosuppressants..)
* affected by any known diseases, infections or recent surgical procedures within 30 days of study initiation.
* knowingly have HIV or Hepatitis
* history of local radiation therapy
* affected by limited mental capacity or language skills such that study information cannot be understood, informed consent cannot be obtained, or simple instructions cannot be followed.
* presented an acute endodontic lesion in the test tooth or in the neighbouring areas to the experimental procedure
* smokers
* suffering from a known psychological disorder

Min Age: 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2015-11

PRIMARY OUTCOMES:
alveolar bone width and height alveolar bone changes in width and height | within 10 days from tooth extraction and at 3 months (+/- 15 days)
  By the use of CBCT scans, alveolar bone changes in width and height will be recorded just after tooth extraction and 3 months later

SECONDARY OUTCOMES:
- Clinical changes of soft and hard tissue and of periodontal parameters in the neighbouring teeth; - Accuracy of panoramic morphometric indexes in detecting osteoporosis | after tooth extraction (once the coagulation has been allowed) and at 3 months (+/- 15 days)
  * By the use of a probe, periodontal parameters in the neighbouring teeth and relevant clinical changes of the alveolar ridge will be recorded
  * On a panoramic radiograph quantitative and qualitative indexes will be calculated and their accuracy in detecting osteoporosis assessed

CONTACTS AND LOCATIONS:
Overall Officials: Nikolaos Donos, Professor, Study Chair — UCL Eastman Dental Institute
Locations (1):
- Eastman Clinical Investigation Centre, London, United Kingdom

REFERENCES:
- [Background] Cortet B. Bone repair in osteoporotic bone: postmenopausal and cortisone-induced osteoporosis. Osteoporos Int. 2011 Jun;22(6):2007-10. doi: 10.1007/s00198-011-1612-3. PMID 21523399
- [Background] Shimizu M, Furuya R, Kawawa T, Sasaki T. Bone wound healing after maxillary molar extraction in ovariectomized aged rats: quantitative backscattered electron image analysis. Anat Rec. 2000 May 1;259(1):76-85. doi: 10.1002/(SICI)1097-0185(20000501)259:13.0.CO;2-0. PMID 10760746
- [Background] Tanaka S, Shimizu M, Debari K, Furuya R, Kawawa T, Sasaki T. Acute effects of ovariectomy on wound healing of alveolar bone after maxillary molar extraction in aged rats. Anat Rec. 2001 Feb 1;262(2):203-12. doi: 10.1002/1097-0185(20010201)262:23.0.CO;2-#. PMID 11169915
- [Background] He YX, Zhang G, Pan XH, Liu Z, Zheng LZ, Chan CW, Lee KM, Cao YP, Li G, Wei L, Hung LK, Leung KS, Qin L. Impaired bone healing pattern in mice with ovariectomy-induced osteoporosis: A drill-hole defect model. Bone. 2011 Jun 1;48(6):1388-400. doi: 10.1016/j.bone.2011.03.720. Epub 2011 Mar 21. PMID 21421090
- [Background] Erdogan O, Shafer DM, Taxel P, Freilich MA. A review of the association between osteoporosis and alveolar ridge augmentation. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2007 Dec;104(6):738.e1-13. doi: 10.1016/j.tripleo.2007.04.008. Epub 2007 Jul 26. PMID 17656117